CLINICAL TRIAL: NCT06592573
Title: Impact of Online or In-person Cognitive Behavioural Psychotherapy Interventions on Anxiety and Depression Symptoms in Caregivers of Patients with Cancer
Brief Title: Online or In-person Interventions on Anxiety and Depression Symptoms in Caregivers of Patients with Cancer
Acronym: CBT_ONLINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione ANT Italia ONLUS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 614-2023-OSS-AUSLBO
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anxiety; Depressive Symptoms
Keywords: Online Psychotherapy; Cargivers; Cancer; Grief; Cognitive-Behavioural Therapy
MeSH Terms: conditions — Anxiety Disorders; Depression; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT_ONLINE (Experimental): 10-12 sessions of cognitive behavioural therapy conducted online.
  Interventions: Other: CBT_ONLINE
- CBT_IN PERSON (Active Comparator): 10-12 sessions of cognitive behavioural therapy conducted in-person.
  Interventions: Other: CBT_IN PERSON

INTERVENTIONS:
Other: CBT_ONLINE — 10-12 sessions of cognitive behavioural therapy conducted online
  Arms: CBT_ONLINE
Other: CBT_IN PERSON — 10-12 sessions of cognitive behavioural therapy conducted in-person.
  Arms: CBT_IN PERSON

SUMMARY:
Oncological diseases are considered a family disease because when one member is diagnosed with cancer, the psycho-physical, social and economic consequences affect the entire family. In Italy, approximately 17% of the population assists a family member. These caregivers are typically unpaid individuals such as partners, offspring, and relatives who provide daily support. In Italy, the prevalence of depressive disorders among caregivers of patients with cancer ranges between 40%-70%. Therefore, providing psychological support to patients and their caregivers throughout the illness and beyond is essential. This support should include the assistance of psychologists and psychotherapists experienced in coping with illness and grieving. Cognitive Behavioral Therapy (CBT) refers to a series of interventions aimed at treating psychological disorders by modifying dysfunctional cognitive factors that sustain and exacerbate this condition. In the telemedicine setting, psychological teleconsultation is experiencing extensive development, especially in the home setting for chronic illnesses. According to the scientific literature, much evidence suggests no difference in the effectiveness of psychological therapies provided telematically or in-person.

This study aims to evaluate the impact of CBT online or in-person intervention on anxiety and depression symptoms. The intervention is designed for caregivers of patients with cancer assisted at home. The sample population consists of caregivers of patients assisted by the oncological palliative home care programme of ANT Foundation and caregivers grieving for a loved one previously assisted by ANT Foundation.

Participants meeting the inclusion criteria will be randomised into two groups:

Online group: caregivers will receive an intervention of 10-12 psychological sessions in the online setting.

In-person group: caregivers will receive the same CBT intervention lasting 10-12 psychological sessions, in-person.

We are expecting:

* Reduction in anxiety symptoms measured by comparison of the results obtained at T0 and T1 of the Generalized Anxiety Disorder Scale-7 (GAD-7) questionnaire
* Reduction in depressive symptoms measured by comparing the results obtained at T0 and T1 of the Patient Health Questionnaire-9 (PHQ-9) questionnaire.

DETAILED DESCRIPTION:
Background Oncological diseases are considered a family disease because when one member is diagnosed with cancer, the psycho-physical, social and economic consequences affect the entire family. In Italy, approximately 17% of the population assists a family member. These caregivers are typically unpaid individuals such as partners, offspring, relatives who provide daily support. In Italy, the prevalence of depressive disorders among caregivers of patients with cancer ranges from 40% to 70%. Providing psychological support to patients and their caregivers throughout the course of the illness, including post-bereavement, is essential This support should include the assistance of psychologists and psychotherapists experienced in coping with illness and grieving.

Cognitive Behavioral Therapy (CBT) refers to a series of interventions aimed at treating psychological disorders by modifying dysfunctional cognitive factors that sustain and exacerbate this condition. In the telemedicine setting, psychological teleconsultation is experiencing extensive development, especially in the home setting for chronic illnesses. Web-based psychological interventions have been proven effective in reducing anxiety and depression symptoms and in improving the quality of life among various patient populations and their relatives. The clinical outcomes are also comparable to psychological interventions delivered in-person. Finally, a great deal of evidence suggests that there is no difference in the effectiveness of psychological therapies provided online or in-person.

Aim of the study The study aims to evaluate the impact of a CBT intervention conducted online or in-person on anxiety and depression symptoms. The intervention is designed for caregivers of patients with cancer assisted at home and for caregivers grieving for a loved one previously assisted at home.

Primary aim

- Evaluation of the impact of a CBT intervention conducted online or in-person on anxiety and depression symptoms.

Secondary aims

* Comparison between the results obtained with CBT intervention delivered online and the same intervention delivered in-person.
* Evaluation of the therapists' degree of familiarity with the online setting.
* Evaluation of the caregivers' degree of satisfaction with the online intervention.

Study setting and target population

The sample population consists of:

i) caregivers of cancer patients assisted by the oncological palliative home care program of ANT Foundation; ii) caregivers grieving for a loved one previously assisted by ANT Foundation. This study model is part of the home care program provided by ANT Foundation which takes care of patients with advanced cancer by focusing not only on the physical effects of the disease but also on the patient's perception of health, with the primary objective of improving quality of life of the patients and families, even after the possible death of sick loved one. ANT Foundation aims to offer the possibility of living the last period of life in one's family environment, acting on pain, suffering and physical and psychological difficulties and on all the complex needs characterizing the end-of-life. Each patient is supported by a multidisciplinary team of physicians, nurses, and psychologists.

Study design The study follows a randomised, drug-free, non-profit, exploratory pre-post interventional design.

Participants meeting the inclusion criteria will be randomized into two groups:

* Online group: caregivers or caregivers in bereavement processing will receive an intervention of 10-12 psychological sessions of CBT in an online setting.
* In-person group: caregivers or caregivers in bereavement processing will receive the same CBT intervention lasting 10-12 sessions, in-person.

If the participant does not have an Internet connection and a tool for tele-consultations, ANT Foundation will provide.

Recruitment and data collection During the first psychological session, the psychologist will explain the study and propose the participation to caregivers. Once consent has been obtained, the psychologist will administer questionnaires to assess anxiety and depression symptoms.

Caregivers meeting the inclusion criteria will be randomized by the ANT Research Department into two arms (Online vs In-person Group) using a series of random numbers generated by Excel.

Randomization The participants will be randomly assigned by the Research Department to online (25 participants) or in-person group (25 participants) by a stratified randomization using a random number list generated by Excel. The randomization list will be kept secret (password protected) from the psychotherapists who will recruit the caregivers. Furthermore, the psychologists will not know to which group the next caregiver will be assigned.

Sample size It is expected that 50 participants will be included. Power analysis The study's power was assessed by considering the reduction of anxiety and depression symptoms (PHQ-9 and CAD-7 questionnaire scores) among 45 caregivers (estimating a 10% dropout) between T0 and T1. The effect size was assumed based on studies in the literature on the effect of a CBT intervention on depression (0.48-0.58) and anxiety (0.38). The power of the study, calculated using G*Power software with a power post hoc analysis for a Wilcoxon test for repeated measures, with α = 0.05, results in (1-β) = 0.68 for an effect size = 0.38, (1-β) = 0.86 for an effect size = 0.48 and (1-β) = 0.96 for an effect size = 0.58. The power of the study for 45 caregivers will range between 0.68 and 0.96.

Psychologists involved in the study Eight psychologists and psychotherapists specialized in Cognitive-Behavioral Therapy (CBT) will participate in the study.

Supervisions and intervisions Monthly and for the entire duration of the study, the psychologists involved in the project will participate in supervision, coordinated by a Cognitive-Behavioural psychotherapist, expert in the management of group dynamics, both in business and health contexts, to manage any issues that emerge during the work. In addition, periodic intervisions will be planned, to promote an exchange on reciprocal intervention experiences acquired during clinical activity, aiming at broadening the frame of observation of problems and solutions and facilitating professionals in the relationship with the patient.

Method The intervention framework is based on the theoretical principles and techniques used in CBT. These therapeutic strategies are designed for targeted and customized interventions for the specific audience of caregivers of cancer patients. To this end, the therapeutic intervention used in the present study is built on the format of Internet-based CBT programs (ICBT) of recognized effectiveness.

The intervention lasts 10-12 psychological sessions and includes a first phase of diagnosis-assessment devoted to case formulation and a second intervention phase devoted to the therapeutic process.The clinical intervention is organized into 11 modules that represent a structural and conceptual guide and must be adapted by the therapist based on the specific needs of the individual caregiver. It is specified that the modules do not coincide with the progressive and sequential steps of therapy but represent a thematic and instrumental guide that the psychologists will refer to. The modules can be overlapping, repeatable and interchangeable depending on the needs that emerge during the course. The aim is to provide a shared and operational structure available to psychologists, but, at the same time, to ensure flexibility and adaptability tailored to the contingency and peculiarities of each case.

Two introductory modules are devoted to the initial psychological sessions and problem analysis:

1. Introduction to the problem.
2. Problem analysis. The goal of the first clinical sessions is to gather basic anamnestic information such as the caregiver's medical and family history, through active and empathic listening aimed at collecting the data necessary for a comprehensive understanding and analysis of the problem. In this way, automatic negative thoughts and core beliefs are identified to arrive at a definition of the therapeutic goals to be shared with the caregiver. The tools that can be used by professionals fall within the range of recognized techniques routinely used in CBT, such as the ABC technique, CEPA Functional Analysis, the Thought Diary, and the Coping Styles Worksheet.

   After the case formulation phase, the subsequent therapeutic process is developed in 8 specific modules plus an additional module on grief divided by objectives:
3. Psycho-education phase: information is shared with the caregiver about the CBT approach according to which the intervention is set up, and in which an attempt is made to increase awareness of the caregiving role and the resulting burden.
4. Changing dysfunctional cognitions: tools such as the Socratic dialogue and cognitive restructuring and reactions on the emotional level are used.
5. Enhancement of coping skills: coping with the changes that illness brings about in daily life.
6. Enhancement of social skills fostering the building and maintenance of support networks.
7. Empowerment of the family member's resources: focus on their specific needs.
8. Acceptance of change and illness of loved one: practices such as mindfulness, ACT, etc. are used.
9. Drafting and planning a series of pleasant activities to lighten the caregiving burden. Tools such as pleasant activity scheduling, relapse prevention plan, etc. are used.
10. Phase of feedback and evaluation of the intervention outcomes: shared verification of the changes and achievement of the set goals, enhancement of the resources that emerged in the therapeutic path to better manage the difficulties identified.
11. Bereavement Processing: in a setting of caring for advanced cancer patients, there is a possibility that the progression of the disease will lead caregivers to confront the death of the family member. Clearly, the caregiver's psychological intake pathway must take this possibility into account and adjust the intervention to include work on possible grief processing. For this purpose, the protocol includes a specific module dedicated to the characteristic challenges of processing loss, within which the therapist can move to restructure goals and adapt them to the contingency of grief, following the cognitive-behavioral Dual Process Model.

The concluding phase is also devoted to assessing the caregiver's satisfaction with the intervention by filling out a dedicated questionnaire at T1.

As mentioned, the therapist will tailor the intervention based on the case formulation and the caregiver's needs and requests, following the structure of the protocol and the specific objectives of each module.

ELIGIBILITY:
Inclusion Criteria:

* Presence of anxious-depressive symptomatology, included in the cut-off 5-21 of the Generalized Anxiety Disorder Scale-7 (GAD-7) and/or in the cut-off 5-27 of the Patient Health Questionnaire-9 (PHQ-9).
* Aged 18 years or older.
* Able to understand the aims of the study and to sign the informed consent.
* Able to understand the Italian language.
* Able to use a technological tool for tele-consultations (smartphone, tablet, computer, etc.).

Exclusion Criteria:

* With severe psychiatric pathology causing clinically significant impairment of functioning in social, occupational or other important areas.
* With cognitive impairment.
* Engaged in psychological support/psychotherapy within the last 3 months.
* Who does not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 for the assessment of depression symptomatology | The questionnaire will be filled out by the participant at the time of recruitment (baseline, T0) and at the end of the intervention (T1, week 13).
  The Patient Health Questionnaire - 9 is the major depressive disorder module of the full questionnaire. This scale is used to provisionally diagnose depression and grade severity of symptoms in general medical and mental health settings. The scores of the 9 questions range from "0" (not at all) to "3" (nearly every day), providing a 0-27 severity total score. The last item ("How difficult have these problems made it for you to do your work, take care of things at home, or get along with other people?") is not included in score, but is a good indicator of the patient's global impairment and can be used to track treatment response. Higher questionnaire scores are associated with decreased functional status and increased symptom-related difficulties, sick days, and healthcare utilization.
Generalized Anxiety Disorder Scale-7 for the assessment of anxiety symptomatology. | The questionnaire will be filled out by the participant at the time of recruitment (baseline, T0) and at the end of the intervention (T1, week 13).
  The General Anxiety Disorder-7 is a rapid screening for the presence of a clinically significant anxiety disorder, especially in outpatient settings. The questionnaire consists of 7 questions and reflects the frequency of symptoms during the preceding 2-week period. The questionnaire requires approximately 1-2 minutes to administer and for each symptom queried provides the following response options: "not at all," "several days," "over half the days" and "nearly every day" and these are scored, respectively, as 0, 1, 2 or 3, providing a 0-21 severity total score. Higher questionnaire scores correlate with disability and functional impairment (in measures such as work productivity and health care utilization).

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Varani, Principal Investigator — Fondazione ANT Italia ONLUS
Locations (1):
- Fondazione ANT, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No